CLINICAL TRIAL: NCT02249663
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multi-Site Study to Evaluate the Therapeutic Equivalence of Azelastine Hydrochloride and Fluticasone Propionate, 137/50 mcg Nasal Spray, to Dymista™ Nasal Spray
Brief Title: Clinical Equivalence of Azelastine Hydrochloride and Fluticasone Propionate, 137/50 mcg Nasal Spray to Dymista™
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 71336006
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Bioequivalence
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Investigational Test Product (Experimental): Azelastine hydrochloride and Fluticasone propionate Nasal Spray, 137/50 mcg
  Interventions: Drug: Azelastine hydrochloride and Fluticasone propionate
- Reference Listed Drug (Active Comparator): Dymista™ (azelastine hydrochloride/fluticasone propionate) Nasal Spray, 137/50 mcg
  Interventions: Drug: Dymista™
- Placebo (Placebo Comparator): Placebo Nasal Spray
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azelastine hydrochloride and Fluticasone propionate — 137/50 mcg Nasal Spray
  Arms: Investigational Test Product
Drug: Dymista™ — 137/50 mcg Nasal Spray
  Other Names: Azelastine hydrochloride and Fluticasone propionate (generic name)
  Arms: Reference Listed Drug
Other: Placebo — Nasal spray with no pharmaceutically active content
  Arms: Placebo

SUMMARY:
To evaluate the therapeutic equivalence of a test formulation of Azelastine hydrochloride and Fluticasone propionate Nasal Spray to the reference listed drug, Dymista™ Nasal Spray in the relief of the signs and symptoms of Seasonal Allergic Rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 12 years of age or older.
* Signed informed consent form, which meets all criteria of current FDA regulations. For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way to be understandable to a child.
* Documented positive allergic skin test, performed within the previous 12 months, to one or more of the allergens in season at the time the study is being conducted.
* A minimum of two consecutive years of previous history of Seasonal Allergic Rhinitis (SAR) to the pollen/allergen in season at the time the study is being conducted.
* Eligibility requirements for placebo lead-in period: A total (composite) score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) with a minimum of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms and total (composite) score of at least 4 on the reflective Total Ocular Symptom Score (rTOSS). These scores represent the 12 hours before the screening visit.
* In addition to requirements above, patients should have the following at the end of the placebo lead-in period and before randomization: 1) average composite score of at least 6 on the rTNSS with a minimum average score of at least 2 for "nasal congestion" and a minimum average score of at least 2 for one of the remaining 3 symptoms, and 2) average composite score of at least 4 on the rTOSS. These scores represent the 3 days of the 7 day placebo run-in period before the Randomization visit and the morning of the first day of the Randomization visit.

Exclusion Criteria:

* Under 12 years of age.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Negative or lack of documented skin allergen test (performed within the previous 12 months) to at least one of the allergens in season at the time the study is being conducted. The results of all positive skin allergen test results should be reported.
* Patients who suffer from chronic signs and symptoms of Perennial Allergic Rhinitis (PAR) should be excluded from the study unless the Investigator assesses that the patient's current signs and symptoms are a clear exacerbation of Seasonal Allergic Rhinitis (SAR) rather than the chronic PAR.
* Patients who suffer only from PAR or SAR to a different allergen than that in season at the time the study is conducted.
* Previous history of less than 2 years of SAR to the pollen/allergen in season at the time the study is conducted.
* Before the placebo lead-in period, the patient has a total score of less than 6 on the rTNSS or a score less than 2 for "nasal congestion". Any patient who meets the minimum individual nasal symptom score requirements at the start of the placebo lead-in period but no longer meets the requirements prior to the randomized active treatment period of the study cannot continue in the active treatment period.
* At the end of the placebo lead-in period and before randomization, the patient has an average composite score of less than 6 on the rTNSS and an average composite score of less than 4 on the rTOSS.
* History of asthma over the previous 2 years that required chronic therapy. Occasional acute or mild exercise induced asthma will be allowable on the condition that the treatment of the attacks is restricted to beta-agonists only.
* Patients with nasal conditions, including infectious rhinitis, rhinitis medicamentosa, or atrophic rhinitis.
* Clinically significant nasal deformity or any recent nasal surgery or trauma that has not completely healed.
* Sinus infection within the previous 30 days or history or re-occurring sinus infections.
* Patient has started immunotherapy or changed their dose of immunotherapy within 30 days of the first placebo lead-in dose or is likely to have to start immunotherapy, or change their current dose during the study.
* Treatment for oral Candidiasis within 30 days of starting the study or a current oral Candidiasis infection.
* Upper respiratory tract infection within the previous 30 days.
* Patients with a history of tuberculosis.
* Patients with presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis, or other eye infection not related to the diagnosis of SAR within 14 days of enrollment.
* The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.
* Patients with any untreated fungal, bacterial, or systemic viral infections within the previous 30 days.
* Use of any ophthalmic steroids within 14 days or nasal, inhaled, or systemic steroids within 30 days of the study start. Super or high potency topical steroids should not be used during the study.
* Use of medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4.
* Use of intranasal or systemic second-generation anti-histamines within 10 days or enrollment.
* Use of intranasal cromolyn within 14 days of enrollment.
* Use of intranasal or systemic first-generation anti-histamines, leukotriene receptor antagonsits or other nasal decongestants within 3 days of enrollment.
* Use of any tricyclic anti-depressant within 30 days of enrollment.
* Patients with attention-deficit disorder being treated with methylphenidate containing products that have not been on a stable regimen for at least the 30 previous days and who cannot remain of the same dose throughout the study.
* Desensitization therapy to the seasonal allergen that is causing the patient's allergic rhinitis within the previous 6 months.
* Previous SAR and/or PAR that has proven unresponsive to steroid therapy.
* Any known hypersensitivity to azelastine hydrochloride, fluticasone propionate, other steroids, or any components of the study nasal spray.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that in the Investigator's opinion would place the patient at undue risk by participating or could jeopardize the integrity of the study evaluations.
* Receipt of any drug as part of a research study within 30 days prior to the first placebo lead-in dose.
* Planned travel outside of the local area for more than 2 consecutive days or 3 days in total, during the patient's participation in the study.
* Previous participation in this study.
* The patient has a history of non-compliance with medication regimens or treatment protocols in previous clinical studies.
* The patient is a member of the investigational study staff or a member of the family of the investigational study staff.
* The patient currently smokes cigarettes, cigars, and/or pipes and is a heavy smoker (for example, on average more than 10 cigarettes per day).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1535 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average AM/PM reflective Total Nasal Symptom Score (rTNSS). | Days 1 to 14

SECONDARY OUTCOMES:
Change from baseline in average instantaneous Total Nasal Symptom Score (iTNSS). | Days 1 to 14
Change from baseline in average reflective Total Ocular Symptom Score (iTOSS). | Days 1 to 14
Change from baseline in average instantaneous Total Ocular Symptom Score (iTOSS). | Days 1 to 14
Onset of Action | 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Darin Brimhall, DO, FACP, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States